CLINICAL TRIAL: NCT02460965
Title: Understanding Hallucinations (Part II) - fMRI and EEG
Brief Title: Understanding Hallucinations (Part II)
Acronym: UH-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Iris Sommer (Other)
Responsible Party: Sponsor-Investigator, Iris Sommer, Prof.Dr., UMC Utrecht
Organization: UMC Utrecht (Other)
Other Study IDs: UH-2
Record Dates: First submitted 2014-02-24; First posted 2015-06-03 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Hallucinations
MeSH Terms: conditions — Hallucinations

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Patients with schizophrenia
- Patients with borderline personality disorder
- Patients with hearing impairment
- Patients with visual loss
- Patients with Parkinson's Disease
- Patients with Alzheimer's Disease
- Patients with dementia with Lewy Bodies
- Healthy participants

SUMMARY:
Rationale: Hallucinations occur in many patients with different kinds of diseases, including psychiatric, neurological and perceptual impairment. The origin of these hallucinations is only partly understood. This prevents correct prediction of treatment response and hampers the development of new, more effective treatment strategies.

Different subtypes of hallucinations resulting from different neuropathology may exist across diagnostic entities, and be responsive to different treatment strategies. Understanding the origin of these subtypes with use of fMRI and EEG can help to make rational treatment decisions on an individual basis and enhance the development of innovative treatment paradigms.

Objective: The primary objective is to find specific abnormalities on resting state fMRI related to the pathophysiology of different subtypes of hallucinations. Secondary objectives are to find EEG connectivity measures that are related to the pathophysiology of different subtypes of hallucinations, reveal correlating patterns of EEG and fMRI that underlie the experience of hallucinations across different disorders, and to examine the frequency of spontaneous synchronized burst activations in auditory and visual cortices using fMRI.

Study design: The investigators intend to examine neural correlates of hallucinations over different disorders using resting state EEG, fMRI and sMRI in an observational study.

Study population: A total of 140 hallucinating patients will be included, 20 of each of the 7 different diagnostic groups. As a control group, 140 non-hallucinating patients with the same disorder of similar severity will be included.

Main study parameters/endpoints: The main study endpoint is the difference in resting state correlates as measured with fMRI between hallucinating and non-hallucinating participants and between hallucinating individuals of different subtypes, namely: connectivity within the DMN and connectivity of the DMN to sensory cortices and the hippocampal-amygdala complex.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participation in the study will entail an MRI scan of 40 minutes and an EEG measurement of 5 minutes. Total visit time, including preparations, will be approximately 2,5 hours. The risks associated with participation and the benefits to the individuals are negligible. The potential benefit to society in the future is considerable if the findings lead to optimization of treatment strategies and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in the phenomenology/cognition study 13-059.
* Belong to one of the diagnostic groups as described above in 4.1.
* Written informed consent

Exclusion Criteria:

* < 18 years of age
* Any contraindication for a 3Tesla MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will consist of 7 different diagnostic categories. Individuals with hallucinations will have to experience at least one episode of hallucinations over the last month. The control group will consist of non-hallucinating individuals who have the same disorder as the hallucinating individuals and are matched group-wise for severity of the disease, medication, age, sex, handedness and education.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Difference in fMRI resting state correlates between hallucinating and non-hallucinating participants and between hallucinating individuals of different subtypes. | Three years
  The main study endpoint is the difference in resting state correlates as measured with fMRI between hallucinating and non-hallucinating participants and between hallucinating individuals of different subtypes, namely: connectivity within the DMN and connectivity of the DMN to sensory cortices and the hippocampal-amygdala complex.

SECONDARY OUTCOMES:
The difference in EEG correlates between hallucinating and non-hallucinating participants and between hallucinating individuals of different subtypes. | Three years
  The differences in EEG spectral analysis, synchronization likelihood, clustering index, path lengths and assortativity between hallucinating and non-hallucinating participants and between hallucinating individuals of different subtypes.
The auditory and visual cortex responsiveness patterns between hallucinating individuals of different subtypes. | Three years
  The frequency of spontaneous synchronized burst activations in auditory and visual cortices

OTHER OUTCOMES:
Cardio-respiratory rhythms to correct for cardio-respiratory processes in the fMRI signal. | Three years
  In order to remove cardiac and respiratory pulsality effects that contaminate BOLD fMRI time series, cardiac signals and respiration will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Iris Sommer, Prof, Dr., Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands